CLINICAL TRIAL: NCT02705313
Title: Expanded Access Protocol for Therapeutic Use of 177Lu-DOTA0-Tyr3-Octreotate in Patients With Inoperable, Somatostatin Receptor Positive, Neuroendocrine Tumors, Progressive Under Somatostatin Analogue Therapy
Brief Title: EAP 177Lu-DOTA0-Tyr3-Octreotate for Inoperable, SSR+, NETs, Progressive Under SSA Tx
Status: Approved for marketing | Type: Expanded Access
Sponsor: Advanced Accelerator Applications (Industry)
Responsible Party: Sponsor
Other Study IDs: AAA-177Lu-03
Record Dates: First submitted 2016-03-07; First posted 2016-03-10 (Estimated); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Neuroendocrine Tumors
Keywords: neuroendocrine tumors; 177Lu-DOTA0-Tyr3-Octreotate; PRRT
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — lutetium Lu 177 dotatate

INTERVENTIONS:
Drug: 177Lu-DOTA0-Tyr3-Octreotate — The treatment regimen consists of 4 administrations of 7.4 GBq (200 mCi) at the date and time of infusion. The recommended interval between two infusions is 8 weeks, which could be extended up to 16 weeks in case of dose modifying toxicity.
  Other Names: Lutathera

SUMMARY:
Advanced Accelerator Applications is currently pursuing marketing approval for 177Lu-DOTA0-Tyr3-Octreotate (Lutathera). This expanded access therapeutic protocol aims to allow patients suffering from inoperable, somatostatin receptor positive, neuroendocrine tumors, progressive under somatostatin analogue therapy to access the investigational product, 177Lu-DOTA0-Tyr3-Octreotate (Lutathera), prior to its commercial availability.

DETAILED DESCRIPTION:
Advanced Accelerator Applications activated in 2012 a multicenter, stratified, open, randomized, comparator-controlled, parallel-group Phase III study comparing treatment with 177Lu-DOTA0-Tyr3-Octreotate to 60 mg Octreotide LAR in patients with inoperable, progressive, somatostatin receptor positive, midgut carcinoid tumors (NETTER-1 trial, EudraCT number 2011-005049-11, IND number 77219).

Clinical studies, including NETTER-1 for which the primary analysis has been conducted, showed clinical evidence of safety and effectiveness to support the expanded access use without any unreasonable potential risks for the patients in the context of the disease to be treated.

In July 2016, the first patient was treated under an Expanded Access Program (EAP) for inoperable, progressive, somatostatin receptor positive, midgut carcinoid tumors.

Compassionate use programs in Europe include pulmonary NETs. In the US, there were many centers with patients with NETs who did not meet the inclusion criteria for the original EAP. In May 2017, Advanced Accelerator Applications inquired with the FDA if amending the inclusion criteria of the original protocol to include all NETs would be permissible.

In June 2017, Advanced Accelerator Applications was able to submit a revision to the original Expanded Access Program's protocol for 177Lu-DOTA0-Tyr3-Octreotate to include neuroendocrine tumors arising from sites other than midgut.

The locations listed below that are participating in the EAP may have received IRB approval for either the original protocol or the new protocol or both. Please, inquire with the Facility Contact as to which protocol is active at their site.

ELIGIBILITY:
Inclusion Criteria:

* Presence of metastasized or locally advanced neuroendocrine tumor, inoperable (curative intent) at enrollment time, and regardless of the origin of the tumor.
* Ki67 index ≤ 20%
* Patients progressive under SSA (any dose) at the time of enrollment
* Target lesions over-expressing somatostatin receptors according to an appropriate imaging method (e.g. 111In-pentetreotide (Octreoscan) imaging or 68Ga-DOTA0-Tyr3-Octreotate (or 68Ga-edotreotide) imaging)

Exclusion Criteria:

* Either serum creatinine >150 μmol/L (>1.7 mg/dL), or creatinine clearance <50 mL/min calculated by the Cockroft Gault method, eventually confirmed by measured creatinine clearance (or measured glomerular filtration rate (GFR) using plasma clearance methods, not gamma camera-based) <50 mL/min (the measured creatinine clearance / GFR is required only as confirmatory exam).
* Hb concentration <5.0 mmol/L (<8.0 g/dL); WBC <2x109/L (2000/mm3); platelets <75x109/L (75x103/mm3).
* Total bilirubin >3 x ULN.
* Serum albumin <3.0 g/dL unless prothrombin time is within the normal range.
* Pregnancy or lactation.
* For female patients of childbearing potential (defined as < 2 years after last menstruation and not surgically sterile) and male patients, who are not surgically sterile or with female partners of childbearing potential: absence of effective, non-hormonal means of contraception (intrauterine contraceptive device, barrier method of contraception in conjunction with spermicidal gel).
* Any surgery, radioembolization, chemoembolization, chemotherapy and radiofrequency ablation within 12 weeks prior to enrollment.
* Interferons, Everolimus (mTOR-inhibitors) or other systemic therapies within 4 weeks prior to enrollment.
* Known brain metastases, unless these metastases have been treated and stabilized.
* Uncontrolled congestive heart failure (NYHA II, III, IV).
* Uncontrolled diabetes mellitus as defined by a fasting blood glucose >2 ULN.
* Any patient receiving treatment with short-acting Octreotide, which cannot be interrupted for 24 h before and 24 h after the administration of 177Lu-DOTA0-Tyr3-Octreotate, or any patient receiving treatment with Octreotide LAR, which cannot be interrupted for at least 4 weeks before the administration of 177Lu-DOTA0-Tyr3-Octreotate, unless the tumor uptake on target lesions is at least as high as normal liver uptake.
* Patients with any other significant medical, psychiatric, or surgical condition, currently uncontrolled by treatment, which may pose a risk to the patient safety
* Prior external beam radiation therapy to more than 25% of the bone marrow.
* Current spontaneous urinary incontinence making impossible the safe administration of the radioactive IMP.
* Other known co-existing malignancies except non-melanoma skin cancer and carcinoma in situ of the uterine cervix, unless definitively treated and with no evidence of recurrence.
* Patients who have not provided a signed informed consent form to accept this treatment.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (41):
- United States (41):
  - Banner M.D. Anderson Cancer Center, Gilbert, Arizona
  - Mayo Clinic Hospital, Phoenix, Arizona
  - City of Hope (City of Hope Medical Center, City of Hope National Medical Center), Duarte, California
  - University of California, Los Angeles, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Kaiser Permanente, Santa Clara Homestead, Santa Clara, California
  - Stanford University Medical Center, Stanford, California
  - University of Colorado Hospital - Anschutz Cancer Pavilion, Aurora, Colorado
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Mayo Clinic, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Cancer Treatment Center of America - Southeastern Regional Medical Center, Newnan, Georgia
  - Northwestern Medicine, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - The University of Iowa Hospitals & Clinics (UIHC) including the Carver College of Medicine, Iowa City, Iowa
  - Ochsner Medical Center, Kenner, Louisiana
  - Johns Hopkins Outpatient Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Kansas City Research Institute, Kansas City, Missouri
  - Washington University School of Medicine Siteman Cancer Center, St Louis, Missouri
  - CHI Health West Omaha Imaging Center, Omaha, Nebraska
  - Roswell Park Cancer Institute, Buffalo, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Stony Brook Cancer Center, Stony Brook, New York
  - Montefiore Einstein Center for Cancer Care, The Bronx, New York
  - Duke University Hospital, Durham, North Carolina
  - The Ohio State University James Cancer Center, Columbus, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh, Medical Center, Pittsburgh, Pennsylvania
  - Bon Secours Medical Group/ Saint Francis Hospital Cancer Center, Greenville, South Carolina
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Utah, Huntsman Cancer Institute, Salt Lake City, Utah
  - Carilion Clinic, Roanoke, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - University of Washington, Department of Radiology, Division of Nuclear Medicine, Seattle, Washington